CLINICAL TRIAL: NCT02218710
Title: Bone Geometry, Volumetric Density, Microarchitecture and Estimated Bone Strength Assessed by High Resolution Peripheral Quantitative Computed Tomography in Patients With Adult Onset Growth Hormone Deficiency
Brief Title: Bone Structure in Patients With Adult Onset Growth Hormone Deficiency Assessed Using High Resolution Peripheral Quantitative Computed Tomography
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Andersen, Associate Professor, DM, DMSc, PhD, Odense University Hospital
Other Study IDs: S-20120156
Record Dates: First submitted 2014-08-07; First posted 2014-08-18 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Adult Onset Growth Hormone Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Growth hormone deficiency (GHD): Pituitary patients with GHD
- healthy controls: Sex and age-matched healthy controls

SUMMARY:
The aim of the study is to assess bone geometry, bone compartment specific volumetric densities and micro-architecture as well as to evaluate non-invasive estimates of bone strength in patients with adult onset growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with Adult onset Growth Hormone Deficiency
* Age between 18-80
* Informed consent

Exclusion Criteria:

* Competing bone disease (e.g.. Mb. Paget, myelomatosis, osteogenesis imperfecta, osteoporosis, primary hyperparathyroidism)
* Ongoing medical treatment affecting bone metabolism (eg. osteoporosis medications)
* Ongoing pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are all seen at the Odense University Hospital at the department of Endocrinology. All patients at the hypophysis clinic were checked and those receiving growth hormone replacement therapy were invited to participate.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
volumetric bone mineral density in grams per cc | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Endocrinological department M, Odense University Hospital, Odense, Region Syddanmark
  - Department M, Odense
  - Department of Endocrinology, Odense University Hospital, Odense